CLINICAL TRIAL: NCT00603512
Title: A Phase 2, Randomized, Double-blind, Placebo-controlled, Multicenter Study to Confirm Dose Responsiveness Following 12 Weeks of the Administration of CP-690,550 (4 Doses) or Placebo in Subjects With Active Rheumatoid Arthritis Inadequately Controlled With Methotrexate Alone
Brief Title: Comparison Of 4 CP-690,550 Doses Vs. Placebo, Each Combined With Methotrexate, For The Treatment Of Rheumatoid Arthritis in Japan
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: A3921039
Record Dates: First submitted 2008-01-17; First posted 2008-01-29 (Estimated); Results first posted 2013-01-25 (Estimated); Last update posted 2013-01-25 (Estimated); Status verified 2012-12

CONDITIONS: Arthritis, Rheumatoid
Keywords: Phase II MTX add-on study in Japan
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — tofacitinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- CP-690,550, 0mg (Placebo Comparator)
  Interventions: Drug: Placebo
- CP-690,550, 10mg (Experimental)
  Interventions: Drug: CP-690,550
- CP-690,550, 1mg (Experimental)
  Interventions: Drug: CP-690,550
- CP-690,550, 3mg (Experimental)
  Interventions: Drug: CP-690,550
- CP-690,550, 5mg (Experimental)
  Interventions: Drug: CP-690,550

INTERVENTIONS:
Drug: Placebo — 0 mg BID, 3 blinded tablets administered BID for 12 weeks
  Arms: CP-690,550, 0mg
Drug: CP-690,550 — 10 mg BID, 3 blinded tablets administered BID for 12 weeks
  Arms: CP-690,550, 10mg
Drug: CP-690,550 — 1 mg BID, 3 blinded tablets administered BID for 12 weeks
  Arms: CP-690,550, 1mg
Drug: CP-690,550 — 3 mg BID, 3 blinded tablets administered BID for 12 weeks
  Arms: CP-690,550, 3mg
Drug: CP-690,550 — 5 mg BID, 3 blinded tablets administered BID for 12 weeks
  Arms: CP-690,550, 5mg

SUMMARY:
The purpose of this study is to determine the effectiveness and safety, over 3 months, of 4 dose regimens of CP-690,550, combined with methotrexate, for the treatment with active rheumatoid arthritis.

ELIGIBILITY:
Inclusion Criteria:

* Active rheumatoid arthritis
* Inadequate response to stably dosed methotrexate

Exclusion Criteria:

* Current therapy with any DMARD or biologic other than methotrexate

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2008-01; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (18):
- Japan (18):
  - Pfizer Investigational Site, Chiba, Chiba
  - Pfizer Investigational Site, Fukuoka, Fukuoka
  - Pfizer Investigational Site, Hitachi-shi, Ibaraki
  - Pfizer Investigational Site, Sagamihara, Kanagawa
  - Pfizer Investigational Site, Yahatanishi-ku, Kitakyusyu
  - Pfizer Investigational Site, Koushi, Kumamoto
  - Pfizer Investigational Site, Sendai, Miyagi
  - Pfizer Investigational Site, Niigata, Niigata
  - Pfizer Investigational Site, Kawachi-Nagano, Osaka
  - Pfizer Investigational Site, Kawagoe-shi, Saitama
  - Pfizer Investigational Site, Kitamoto, Saitama
  - Pfizer Investigational Site, Bunkyo-ku, Tokyo
  - Pfizer Investigational Site, Bunkyo-k, Tokyo
  - Pfizer Investigational Site, Chiyoda-ku, Tokyo
  - Pfizer Investigational Site, Koto-ku, Tokyo
  - Pfizer Investigational Site, Meguro-ku, Tokyo
  - Pfizer Investigational Site, Musashimurayama-shi, Tokyo
  - Pfizer Investigational Site, Shinjyuku-ku, Tokyo

REFERENCES:
- [Derived] Hetland ML, Strangfeld A, Bonfanti G, Soudis D, Deuring JJ, Edwards RA. Machine learning prediction and explanatory models of serious infections in patients with rheumatoid arthritis treated with tofacitinib. Arthritis Res Ther. 2024 Aug 27;26(1):153. doi: 10.1186/s13075-024-03376-9. PMID 39192350
- [Derived] Wright GC, Mysler E, Kwok K, Cadatal MJ, Germino R, Yndestad A, Kinch CD, Ogdie A. Impact of Race on the Efficacy and Safety of Tofacitinib in Rheumatoid Arthritis: Post Hoc Analysis of Pooled Clinical Trials. Rheumatol Ther. 2024 Oct;11(5):1135-1164. doi: 10.1007/s40744-024-00677-y. Epub 2024 Jul 3. PMID 38958913
- [Derived] Kristensen LE, Danese S, Yndestad A, Wang C, Nagy E, Modesto I, Rivas J, Benda B. Identification of two tofacitinib subpopulations with different relative risk versus TNF inhibitors: an analysis of the open label, randomised controlled study ORAL Surveillance. Ann Rheum Dis. 2023 Jul;82(7):901-910. doi: 10.1136/ard-2022-223715. Epub 2023 Mar 17. PMID 36931693
- [Derived] Hansen KE, Mortezavi M, Nagy E, Wang C, Connell CA, Radi Z, Litman HJ, Adami G, Rossini M. Fracture in clinical studies of tofacitinib in rheumatoid arthritis. Ther Adv Musculoskelet Dis. 2022 Dec 27;14:1759720X221142346. doi: 10.1177/1759720X221142346. eCollection 2022. PMID 36601090
- [Derived] Curtis JR, Yamaoka K, Chen YH, Bhatt DL, Gunay LM, Sugiyama N, Connell CA, Wang C, Wu J, Menon S, Vranic I, Gomez-Reino JJ. Malignancy risk with tofacitinib versus TNF inhibitors in rheumatoid arthritis: results from the open-label, randomised controlled ORAL Surveillance trial. Ann Rheum Dis. 2023 Mar;82(3):331-343. doi: 10.1136/ard-2022-222543. Epub 2022 Dec 5. PMID 36600185
- [Derived] Winthrop KL, Yndestad A, Henrohn D, Danese S, Marsal S, Galindo M, Woolcott JC, Jo H, Kwok K, Shapiro AB, Jones TV, Diehl A, Su C, Panes J, Cohen SB. Influenza Adverse Events in Patients with Rheumatoid Arthritis, Ulcerative Colitis, or Psoriatic Arthritis in the Tofacitinib Clinical Development Programs. Rheumatol Ther. 2023 Apr;10(2):357-373. doi: 10.1007/s40744-022-00507-z. Epub 2022 Dec 17. PMID 36526796
- [Derived] Winthrop KL, Curtis JR, Yamaoka K, Lee EB, Hirose T, Rivas JL, Kwok K, Burmester GR. Clinical Management of Herpes Zoster in Patients With Rheumatoid Arthritis or Psoriatic Arthritis Receiving Tofacitinib Treatment. Rheumatol Ther. 2022 Feb;9(1):243-263. doi: 10.1007/s40744-021-00390-0. Epub 2021 Dec 6. PMID 34870800
- [Derived] Cohen SB, Tanaka Y, Mariette X, Curtis JR, Lee EB, Nash P, Winthrop KL, Charles-Schoeman C, Wang L, Chen C, Kwok K, Biswas P, Shapiro A, Madsen A, Wollenhaupt J. Long-term safety of tofacitinib up to 9.5 years: a comprehensive integrated analysis of the rheumatoid arthritis clinical development programme. RMD Open. 2020 Oct;6(3):e001395. doi: 10.1136/rmdopen-2020-001395. PMID 33127856
- [Derived] Panaccione R, Isaacs JD, Chen LA, Wang W, Marren A, Kwok K, Wang L, Chan G, Su C. Characterization of Creatine Kinase Levels in Tofacitinib-Treated Patients with Ulcerative Colitis: Results from Clinical Trials. Dig Dis Sci. 2021 Aug;66(8):2732-2743. doi: 10.1007/s10620-020-06560-4. Epub 2020 Aug 20. PMID 32816215
- [Derived] Mariette X, Chen C, Biswas P, Kwok K, Boy MG. Lymphoma in the Tofacitinib Rheumatoid Arthritis Clinical Development Program. Arthritis Care Res (Hoboken). 2018 May;70(5):685-694. doi: 10.1002/acr.23421. Epub 2018 Apr 2. PMID 28941219
- [Derived] Cohen SB, Tanaka Y, Mariette X, Curtis JR, Lee EB, Nash P, Winthrop KL, Charles-Schoeman C, Thirunavukkarasu K, DeMasi R, Geier J, Kwok K, Wang L, Riese R, Wollenhaupt J. Long-term safety of tofacitinib for the treatment of rheumatoid arthritis up to 8.5 years: integrated analysis of data from the global clinical trials. Ann Rheum Dis. 2017 Jul;76(7):1253-1262. doi: 10.1136/annrheumdis-2016-210457. Epub 2017 Jan 31. PMID 28143815
- [Derived] Charles-Schoeman C, Burmester G, Nash P, Zerbini CA, Soma K, Kwok K, Hendrikx T, Bananis E, Fleischmann R. Efficacy and safety of tofacitinib following inadequate response to conventional synthetic or biological disease-modifying antirheumatic drugs. Ann Rheum Dis. 2016 Jul;75(7):1293-301. doi: 10.1136/annrheumdis-2014-207178. Epub 2015 Aug 14. PMID 26275429
- [Derived] Cohen S, Radominski SC, Gomez-Reino JJ, Wang L, Krishnaswami S, Wood SP, Soma K, Nduaka CI, Kwok K, Valdez H, Benda B, Riese R. Analysis of infections and all-cause mortality in phase II, phase III, and long-term extension studies of tofacitinib in patients with rheumatoid arthritis. Arthritis Rheumatol. 2014 Nov;66(11):2924-37. doi: 10.1002/art.38779. PMID 25047021

RESULTS

PARTICIPANT FLOW:
Groups:
- CP-690,550 1 mg: CP-690,550 1 milligram (mg) tablet orally twice daily for 12 weeks.
- CP-690,550 3 mg: CP-690,550 3 mg tablet orally twice daily for 12 weeks.
- CP-690,550 5 mg: CP-690,550 5 mg tablet orally twice daily for 12 weeks.
- CP-690,550 10 mg: CP-690,550 10 mg tablet orally twice daily for 12 weeks.
- Placebo: Placebo tablet matched to CP-690,550 orally twice daily for 12 weeks.
Period: Overall Study
Arm/Group | CP-690,550 1 mg | CP-690,550 3 mg | CP-690,550 5 mg | CP-690,550 10 mg | Placebo
Started | 28 | 28 | 28 | 28 | 28
Treated | 28 | 27 | 27 | 26 | 28
Completed | 26 | 23 | 23 | 21 | 23
Not Completed | 2 | 5 | 5 | 7 | 5
Not completed — Adverse Event | 0 | 2 | 4 | 4 | 2
Not completed — Lack of Efficacy | 0 | 1 | 0 | 0 | 1
Not completed — Other | 2 | 1 | 0 | 1 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 1
Not completed — Randomized but not treated | 0 | 1 | 1 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CP-690,550 1 mg | CP-690,550 3 mg | CP-690,550 5 mg | CP-690,550 10 mg | Placebo | Total
Number analyzed (Participants) | 28 | 27 | 27 | 26 | 28 | 136
Age Continuous [Mean (Standard Deviation); unit: Years] | 52.0 (9.4) | 53.3 (12.1) | 50.0 (9.8) | 50.6 (10.0) | 50.6 (12.4) | 51.3 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 24 | 22 | 25 | 25 | 117
  Male | 7 | 3 | 5 | 1 | 3 | 19

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving American College of Rheumatology 20% (ACR20) Response at Week 12
Description: ACR20 response: greater than or equal to (>=) 20 percent (%) improvement in tender joint count (TJC); >= 20% improvement in swollen joint count (SJC); and >= 20% improvement in at least 3 of 5 remaining ACR core measures: participant assessment of pain; participant global assessment of disease activity; physician global assessment of disease activity; self-assessed disability (disability index of the Health Assessment Questionnaire [HAQ]); and C-Reactive Protein (CRP).
Time Frame: Week 12
Population: Full analysis set (FAS) included all randomized participants who received at least 1 dose of study medication. Missing values were imputed using Last observation carried forward (LOCF) method.
Measure: Number; unit: Percentage of Participants
Arm/Group | CP-690,550 1 mg | CP-690,550 3 mg | CP-690,550 5 mg | CP-690,550 10 mg | Placebo
Number analyzed (Participants) | 28 | 27 | 27 | 26 | 28
Percentage of Participants | 64.3 | 77.8 | 96.3 | 80.8 | 14.3

2. Secondary Outcome: Percentage of Participants Achieving American College of Rheumatology 20% (ACR20) Response
Description: ACR20 response: >= 20% improvement in TJC; >= 20% improvement in SJC; and >= 20% improvement in at least 3 of 5 remaining ACR core measures: participant assessment of pain; participant global assessment of disease activity; physician global assessment of disease activity; self-assessed disability (disability index of the HAQ); and CRP.
Time Frame: Week 1, 2, 4, 8
Population: FAS included all randomized participants who received at least 1 dose of study medication. Missing values were imputed using LOCF method.
Measure: Number; unit: Percentage of Participants
Arm/Group | CP-690,550 1 mg | CP-690,550 3 mg | CP-690,550 5 mg | CP-690,550 10 mg | Placebo
Number analyzed (Participants) | 28 | 27 | 27 | 26 | 28
Percentage of Participants
  Week 1 | 28.57 | 14.81 | 29.63 | 38.46 | 3.57
  Week 2 | 32.14 | 40.74 | 62.96 | 50.00 | 10.71
  Week 4 | 50.00 | 55.56 | 88.89 | 76.92 | 10.71
  Week 8 | 67.86 | 66.67 | 96.30 | 80.77 | 21.43

3. Secondary Outcome: Percentage of Participants Achieving American College of Rheumatology 50% (ACR50) Response
Description: ACR50 response: >= 50% improvement in tender or swollen joint counts and 50% improvement in at least 3 of 5 remaining ACR core measures: participant assessment of pain; participant global assessment of disease activity; physician global assessment of disease activity; self-assessed disability (disability index of the HAQ); and CRP.
Time Frame: Week 1, 2, 4, 8, 12/End of Treatment (EOT)
Population: as for outcome 2
Measure: Number; unit: Percentage of Participants
Arm/Group | CP-690,550 1 mg | CP-690,550 3 mg | CP-690,550 5 mg | CP-690,550 10 mg | Placebo
Number analyzed (Participants) | 28 | 27 | 27 | 26 | 28
Percentage of Participants
  Week 1 | 7.14 | 3.70 | 0.00 | 7.69 | 0.00
  Week 2 | 7.14 | 7.41 | 25.93 | 26.92 | 0.00
  Week 4 | 10.71 | 22.22 | 29.63 | 34.62 | 3.57
  Week 8 | 28.57 | 29.63 | 70.37 | 50.00 | 7.14
  Week 12 | 32.14 | 44.44 | 81.48 | 57.69 | 14.29

4. Secondary Outcome: Percentage of Participants Achieving American College of Rheumatology 70% (ACR70) Response
Description: ACR70 response: >= 70% improvement in tender or swollen joint counts and 70% improvement in at least 3 of 5 remaining ACR core measures: participant assessment of pain; participant global assessment of disease activity; physician global assessment of disease activity; self-assessed disability (disability index of the HAQ); and CRP.
Time Frame: Week 1, 2, 4, 8, 12/EOT
Population: as for outcome 2
Measure: Number; unit: Percentage of Participants
Arm/Group | CP-690,550 1 mg | CP-690,550 3 mg | CP-690,550 5 mg | CP-690,550 10 mg | Placebo
Number analyzed (Participants) | 28 | 27 | 27 | 26 | 28
Percentage of Participants
  Week 1 | 0.00 | 0.00 | 0.00 | 3.85 | 0.00
  Week 2 | 0.00 | 3.70 | 11.11 | 3.85 | 0.00
  Week 4 | 3.57 | 7.41 | 14.81 | 7.69 | 0.00
  Week 8 | 3.57 | 7.41 | 33.33 | 26.92 | 3.57
  Week 12 | 7.14 | 14.81 | 33.33 | 34.62 | 3.57

5. Secondary Outcome: Percentage of Participants Achieving American College of Rheumatology 90% (ACR90) Response
Description: ACR90 response: >= 90% improvement in tender or swollen joint counts and 90% improvement in at least 3 of 5 remaining ACR core measures: participant assessment of pain; participant global assessment of disease activity; physician global assessment of disease activity; self-assessed disability (disability index of the HAQ); and CRP.
Time Frame: Week 1, 2, 4, 8, 12/EOT
Population: as for outcome 2
Measure: Number; unit: Percentage of Participants
Arm/Group | CP-690,550 1 mg | CP-690,550 3 mg | CP-690,550 5 mg | CP-690,550 10 mg | Placebo
Number analyzed (Participants) | 28 | 27 | 27 | 26 | 28
Percentage of Participants
  Week 1 | 0.00 | 0.00 | 0.00 | 0.00 | 0.00
  Week 2 | 0.00 | 0.00 | 0.00 | 3.85 | 0.00
  Week 4 | 0.00 | 0.00 | 3.70 | 0.00 | 0.00
  Week 8 | 0.00 | 3.70 | 7.41 | 3.85 | 0.00
  Week 12 | 0.00 | 11.11 | 3.70 | 11.54 | 0.00

6. Secondary Outcome: Tender Joint Count (TJC)
Description: Number of tender joints was determined by examining 68 joints and identified the joints that were painful under pressure or to passive motion. The number of tender joints was recorded on the joint assessment form at each visit, no tenderness = 0, tenderness = 1.
Time Frame: Baseline, Week 1, 2, 4, 8, 12/EOT
Population: FAS included all randomized participants who received at least 1 dose of study medication. 'n' = number of participants who were evaluable at specific time points for each arm group, respectively.
Measure: Mean (Standard Deviation); unit: tender joints
Arm/Group | CP-690,550 1 mg | CP-690,550 3 mg | CP-690,550 5 mg | CP-690,550 10 mg | Placebo
Number analyzed (Participants) | 28 | 27 | 27 | 26 | 28
tender joints
  Baseline (n=28,27,27,26,28) | 16.36 (7.56) | 16.22 (8.50) | 17.81 (12.32) | 15.42 (9.77) | 16.36 (9.08)
  Week 1 (n=28,26,27,26,28) | 11.89 (7.06) | 12.04 (10.95) | 13.22 (14.04) | 10.96 (11.89) | 12.86 (9.03)
  Week 2 (n=27,27,27,25,26) | 11.63 (8.72) | 9.63 (8.72) | 9.52 (13.12) | 8.20 (10.91) | 11.62 (9.43)
  Week 4 (n=27,26,27,24,25) | 10.04 (7.64) | 7.00 (7.61) | 8.22 (10.48) | 5.58 (6.35) | 13.76 (11.30)
  Week 8 (n=26,25,26,23,24) | 6.73 (6.80) | 5.40 (7.64) | 5.15 (6.49) | 3.35 (4.71) | 11.04 (8.38)
  Week 12 (n=26,24,24,21,24) | 5.92 (6.73) | 6.38 (9.60) | 3.63 (4.39) | 2.71 (4.33) | 9.96 (7.85)

7. Secondary Outcome: Change From Baseline in Tender Joint Count (TJC) at Week 1, 2, 4, 8 and 12/EOT
Description: Number of tender joints was determined by examining 68 joints and identified the joints that were painful under pressure or to passive motion. The number of tender joints was recorded on the joint assessment form at each visit, no tenderness = 0, tenderness = 1. A negative value in change from baseline indicates an improvement.
Time Frame: Baseline, Week 1, 2, 4, 8, 12/EOT
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: tender joints
Arm/Group | CP-690,550 1 mg | CP-690,550 3 mg | CP-690,550 5 mg | CP-690,550 10 mg | Placebo
Number analyzed (Participants) | 28 | 27 | 27 | 26 | 28
tender joints
  Week 1 (n=28,26,27,26,28) | -4.46 (4.80) | -4.19 (6.92) | -4.59 (5.76) | -4.46 (7.61) | -3.50 (5.68)
  Week 2 (n=27,27,27,25,26) | -4.70 (7.37) | -6.59 (7.31) | -8.30 (6.36) | -6.88 (6.09) | -4.54 (5.48)
  Week 4 (n=27,26,27,24,25) | -6.30 (8.78) | -9.00 (8.94) | -9.59 (7.00) | -9.88 (7.50) | -2.28 (8.38)
  Week 8 (n=26,25,26,23,24) | -9.42 (8.90) | -10.84 (9.00) | -12.88 (10.77) | -12.09 (8.23) | -4.04 (7.17)
  Week 12 (n=26,24,24,21,24) | -10.23 (8.84) | -9.96 (10.79) | -14.42 (10.43) | -12.71 (8.01) | -5.13 (7.27)

8. Secondary Outcome: Swollen Joint Count (SJC)
Description: Number of swollen joints was determined by examination of 66 joints and identifying when swelling was present. The number of swollen joints was recorded on the joint assessment form at each visit, no swelling = 0, swelling =1.
Time Frame: Baseline, Week 1, 2, 4, 8, 12/EOT
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: swollen joints
Arm/Group | CP-690,550 1 mg | CP-690,550 3 mg | CP-690,550 5 mg | CP-690,550 10 mg | Placebo
Number analyzed (Participants) | 28 | 27 | 27 | 26 | 28
swollen joints
  Baseline (n=28,27,27,26,28) | 13.18 (5.63) | 15.11 (7.92) | 15.59 (12.41) | 15.12 (9.96) | 13.82 (6.27)
  Week 1 (n=28,26,27,26,28) | 10.07 (5.87) | 12.62 (9.21) | 12.70 (12.66) | 9.73 (10.98) | 13.18 (7.45)
  Week 2 (n=27,27,27,25,26) | 8.26 (4.81) | 9.67 (6.23) | 9.41 (11.52) | 8.04 (11.36) | 12.04 (6.95)
  Week 4 (n=27,26,27,24,25) | 7.85 (6.00) | 8.19 (6.50) | 7.41 (9.28) | 6.63 (7.83) | 11.80 (7.88)
  Week 8 (n=26,25,26,23,24) | 5.92 (4.86) | 6.12 (5.40) | 4.62 (4.99) | 5.17 (6.31) | 11.08 (8.10)
  Week 12 (n=26,24,24,21,24) | 5.19 (5.87) | 5.29 (5.43) | 3.83 (4.24) | 4.05 (5.98) | 11.13 (7.12)

9. Secondary Outcome: Change From Baseline in Swollen Joint Count (SJC) at Week 1, 2, 4, 8 and 12/EOT
Description: Number of swollen joints was determined by examination of 66 joints and identifying when swelling was present. The number of swollen joints was recorded on the joint assessment form at each visit, no swelling = 0, swelling =1. A negative value in change from baseline indicates an improvement.
Time Frame: Baseline, Week 1, 2, 4, 8, 12/EOT
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: swollen joints
Arm/Group | CP-690,550 1 mg | CP-690,550 3 mg | CP-690,550 5 mg | CP-690,550 10 mg | Placebo
Number analyzed (Participants) | 28 | 27 | 27 | 26 | 28
swollen joints
  Week 1 (n=28,26,27,26,28) | -3.11 (5.26) | -2.54 (6.11) | -2.89 (2.81) | -5.38 (5.08) | -0.64 (3.71)
  Week 2 (n=27,27,27,25,26) | -4.74 (5.45) | -5.44 (6.57) | -6.19 (5.02) | -6.84 (4.87) | -1.69 (3.48)
  Week 4 (n=27,26,27,24,25) | -5.15 (7.25) | -6.69 (7.07) | -8.19 (5.94) | -8.50 (5.16) | -1.68 (4.59)
  Week 8 (n=26,25,26,23,24) | -6.92 (6.56) | -8.96 (8.25) | -11.35 (8.91) | -10.09 (6.08) | -2.08 (6.55)
  Week 12 (n=26,24,24,21,24) | -7.65 (7.53) | -9.71 (8.16) | -12.58 (10.06) | -11.71 (6.68) | -2.04 (5.77)

10. Secondary Outcome: Patient Assessment of Arthritis Pain
Description: Participants rated the severity of arthritis pain on a 0 to 100 millimeter (mm) Visual Analog Scale (VAS), where 0 = no pain and 100 = most severe pain.
Time Frame: Baseline, Week 1, 2, 4, 8, 12/EOT
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | CP-690,550 1 mg | CP-690,550 3 mg | CP-690,550 5 mg | CP-690,550 10 mg | Placebo
Number analyzed (Participants) | 28 | 27 | 27 | 26 | 28
mm
  Baseline (n=28,26,27,26,28) | 54.18 (23.48) | 57.59 (20.18) | 53.22 (25.94) | 52.19 (24.97) | 53.32 (23.63)
  Week 1 (n=28,26,27,26,28) | 45.36 (20.32) | 43.50 (20.69) | 40.19 (24.03) | 37.08 (23.38) | 49.36 (24.42)
  Week 2 (n=27,27,27,25,26) | 45.11 (20.11) | 40.52 (24.32) | 33.19 (24.63) | 31.40 (20.92) | 48.58 (25.56)
  Week 4 (n=27,26,27,25,26) | 42.44 (20.98) | 34.88 (22.45) | 25.19 (20.67) | 30.46 (23.60) | 49.72 (24.46)
  Week 8 (n=26,25,27,23,24) | 32.65 (17.84) | 30.04 (23.37) | 22.59 (21.45) | 19.43 (18.64) | 48.88 (23.01)
  Week 12 (n=26,24,24,21,24) | 32.19 (17.69) | 27.17 (21.40) | 17.58 (17.27) | 16.90 (20.29) | 44.96 (25.41)

11. Secondary Outcome: Change From Baseline in Patient Assessment of Arthritis Pain at Week 1, 2, 4, 8 and 12/EOT
Description: Participants rated the severity of arthritis pain on a 0 to 100 mm VAS, where 0 = no pain and 100 = most severe pain.
Time Frame: Baseline, Week 1, 2, 4, 8, 12/EOT
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | CP-690,550 1 mg | CP-690,550 3 mg | CP-690,550 5 mg | CP-690,550 10 mg | Placebo
Number analyzed (Participants) | 28 | 27 | 27 | 26 | 28
mm
  Week 1 (n=28,26,27,26,28) | -8.82 (18.21) | -14.35 (16.99) | -13.04 (18.78) | -15.12 (19.89) | -3.96 (14.90)
  Week 2 n=27,27,27,25,26) | -10.41 (20.16) | -17.07 (25.47) | -20.04 (22.04) | -22.44 (27.77) | -3.69 (10.60)
  Week 4 (n=27,26,27,24,25) | -13.07 (23.22) | -23.35 (22.89) | -28.04 (23.74) | -24.29 (26.28) | -1.00 (14.27)
  Week 8 (n=26,25,27,23,24) | -22.54 (26.84) | -28.92 (23.46) | -30.63 (25.40) | -34.26 (26.19) | -2.04 (22.66)
  Week 12 (n=26,24,24,21,24) | -23.00 (25.13) | -32.50 (22.75) | -31.38 (22.67) | -38.43 (28.38) | -5.96 (22.61)

12. Secondary Outcome: Patient Global Assessment (PtGA) of Arthritis
Description: Participants answered: "Considering all the ways your arthritis affects you, how are you feeling today?" Participants responded by using a 0 - 100 mm VAS, where 0 = very well and 100 = very poorly.
Time Frame: Baseline, Week 1, 2, 4, 8, 12/EOT
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | CP-690,550 1 mg | CP-690,550 3 mg | CP-690,550 5 mg | CP-690,550 10 mg | Placebo
Number analyzed (Participants) | 28 | 27 | 27 | 26 | 28
mm
  Baseline (n=28,27,27,26,28) | 58.00 (18.27) | 60.26 (21.79) | 58.67 (23.63) | 52.04 (26.27) | 53.50 (24.04)
  Week 1 (n=28,26,27,26,28) | 45.89 (21.08) | 44.27 (19.25) | 42.56 (24.48) | 34.73 (21.41) | 46.54 (23.49)
  Week 2 (n=27,27,27,25,26) | 46.07 (22.39) | 42.63 (23.82) | 33.78 (25.04) | 30.44 (20.57) | 48.42 (25.65)
  Week 4 (n=27,26,27,24,25) | 44.59 (22.89) | 34.23 (21.81) | 28.93 (21.61) | 30.04 (22.62) | 49.16 (25.09)
  Week 8 (n=26,25,27,23,24) | 35.12 (17.80) | 30.68 (24.36) | 21.81 (22.22) | 20.39 (20.85) | 49.17 (22.00)
  Week 12 (n=26,24,24,21,24) | 31.42 (17.08) | 24.21 (19.82) | 17.13 (16.00) | 16.48 (18.62) | 43.75 (24.60)

13. Secondary Outcome: Change From Baseline in Patient Global Assessment of Arthritis (PtGA) at Week 1, 2, 4, 8 and 12/EOT
Description: as for outcome 12
Time Frame: Baseline, Week 1, 2, 4, 8, 12/EOT
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | CP-690,550 1 mg | CP-690,550 3 mg | CP-690,550 5 mg | CP-690,550 10 mg | Placebo
Number analyzed (Participants) | 28 | 27 | 27 | 26 | 28
mm
  Week 1 (n=28,26,27,26,28) | -12.11 (17.07) | -16.92 (17.48) | -16.11 (20.72) | -17.31 (20.45) | -6.96 (15.78)
  Week 2 (n=27,27,27,25,26) | -12.19 (18.44) | -17.63 (25.30) | -24.89 (21.03) | -23.40 (28.28) | -3.69 (12.29)
  Week 4 (n=27,26,27,24,25) | -13.67 (20.21) | -27.50 (21.80) | -29.74 (21.90) | -24.50 (26.24) | -1.40 (14.92)
  Week 8 (n=26,25,27,23,24) | -22.85 (25.79) | -32.04 (22.17) | -36.85 (22.07) | -33.09 (27.70) | -1.46 (23.75)
  Week 12 (n=26,24,24,21,24) | -26.54 (24.18) | -38.00 (21.09) | -37.46 (19.91) | -38.33 (29.46) | -6.88 (21.45)

14. Secondary Outcome: Physician Global Assessment (PGA) of Arthritis
Description: Physician Global Assessment of Arthritis was measured on a 0 to 100 mm VAS, where 0 = very good and 100 = very bad.
Time Frame: Baseline, Week 1, 2, 4, 8, 12/EOT
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | CP-690,550 1 mg | CP-690,550 3 mg | CP-690,550 5 mg | CP-690,550 10 mg | Placebo
Number analyzed (Participants) | 28 | 27 | 27 | 26 | 28
mm
  Baseline (n=28,27,27,26,28) | 66.00 (16.32) | 61.44 (19.18) | 59.37 (17.67) | 59.04 (18.00) | 59.39 (19.88)
  Week 1 (n=28,26,27,26,28) | 49.96 (17.44) | 47.96 (19.95) | 45.26 (21.43) | 36.12 (19.45) | 50.64 (22.39)
  Week 2 (n=27,27,27,25,26) | 44.04 (18.74) | 42.52 (23.78) | 34.59 (22.64) | 28.84 (18.90) | 44.62 (22.26)
  Week 4 (n=27,26,27,24,25) | 41.30 (20.94) | 33.04 (18.66) | 24.67 (17.67) | 23.92 (16.60) | 47.96 (23.20)
  Week 8 (n=26,25,26,23,24) | 29.65 (15.94) | 26.08 (18.70) | 17.46 (14.83) | 16.57 (13.62) | 40.21 (21.40)
  Week 12 (n=26,24,24,21,24) | 26.31 (20.39) | 23.38 (17.00) | 13.71 (10.58) | 14.86 (12.28) | 40.92 (21.69)

15. Secondary Outcome: Change From Baseline in Physician Global Assessment of Arthritis (PGA) at Week 1, 2, 4, 8 and 12/EOT
Description: Physician Global Assessment of Arthritis was measured on a 0 to 100 mm VAS, where 0 = very good and 100 = very bad.
Time Frame: Baseline, Week 1, 2, 4, 8, 12/EOT
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | CP-690,550 1 mg | CP-690,550 3 mg | CP-690,550 5 mg | CP-690,550 10 mg | Placebo
Number analyzed (Participants) | 28 | 27 | 27 | 26 | 28
mm
  Week 1 (n=28,26,27,26,28) | -16.04 (15.29) | -14.12 (13.11) | -14.11 (12.67) | -22.92 (21.00) | -8.75 (15.39)
  Week 2 (n=27,27,27,25,26) | -22.33 (18.70) | -18.93 (18.12) | -24.78 (16.65) | -30.16 (20.74) | -13.69 (18.05)
  Week 4 (n=27,26,27,24,25) | -25.07 (25.23) | -28.23 (17.91) | -34.70 (18.49) | -34.83 (19.77) | -9.36 (20.67)
  Week 8 (n=26,25,26,23,24) | -35.88 (23.06) | -35.72 (15.68) | -41.46 (17.19) | -42.17 (19.26) | -16.63 (23.24)
  Week 12 (n=26,24,24,21,24) | -39.23 (27.72) | -36.92 (17.53) | -44.71 (15.94) | -45.05 (20.37) | -15.92 (24.95)

16. Secondary Outcome: Health Assessment Questionnaire-Disability Index (HAQ-DI)
Description: HAQ-DI: participant-reported assessment of ability to perform tasks in 8 categories of daily living activities: dress/groom; arise; eat; walk; reach; grip; hygiene; and common activities over past week. Each item scored on 4-point scale from 0 to 3: 0=no difficulty; 1=some difficulty; 2=much difficulty; 3=unable to do. Overall score was computed as the sum of domain scores and divided by the number of domains answered. Total possible score range 0-3 where 0 = least difficulty and 3 = extreme difficulty.
Time Frame: Baseline, Week 1, 2, 4, 8, 12/EOT
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CP-690,550 1 mg | CP-690,550 3 mg | CP-690,550 5 mg | CP-690,550 10 mg | Placebo
Number analyzed (Participants) | 28 | 27 | 27 | 26 | 28
units on a scale
  Baseline (n=28,27,27,26,28) | 1.14 (0.74) | 1.29 (0.64) | 1.17 (0.60) | 1.16 (0.58) | 1.25 (0.70)
  Week 1 (n=28,26,27,26,28) | 1.05 (0.75) | 1.23 (0.66) | 1.05 (0.54) | 0.85 (0.54) | 1.25 (0.74)
  Week 2 (n=27,27,27,25,26) | 1.04 (0.72) | 1.12 (0.66) | 0.88 (0.56) | 0.79 (0.50) | 1.18 (0.76)
  Week 4 (n=27,26,27,24,25) | 0.94 (0.74) | 1.04 (0.75) | 0.79 (0.55) | 0.77 (0.58) | 1.07 (0.70)
  Week 8 (n=26,25,27,23,24) | 0.80 (0.69) | 0.96 (0.78) | 0.72 (0.54) | 0.64 (0.53) | 1.21 (0.80)
  Week 12 (n=26,24,24,21,24) | 0.78 (0.70) | 0.81 (0.73) | 0.56 (0.41) | 0.59 (0.54) | 1.13 (0.79)

17. Secondary Outcome: Change From Baseline in Health Assessment Questionnaire-Disability Index (HAQ-DI) at Week 1, 2, 4, 8 and 12/EOT
Description: as for outcome 16
Time Frame: Baseline, Week 1, 2, 4, 8, 12/EOT
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CP-690,550 1 mg | CP-690,550 3 mg | CP-690,550 5 mg | CP-690,550 10 mg | Placebo
Number analyzed (Participants) | 28 | 27 | 27 | 26 | 28
units on a scale
  Week 1 (n=28,26,27,26,28) | -0.08 (0.29) | -0.11 (0.37) | -0.12 (0.18) | -0.31 (0.39) | -0.00 (0.19)
  Week 2 (n=27,27,27,25,26) | -0.13 (0.35) | -0.17 (0.39) | -0.29 (0.32) | -0.39 (0.38) | -0.02 (0.26)
  Week 4 (n=27,26,27,24,25) | -0.22 (0.48) | -0.25 (0.47) | -0.38 (0.30) | -0.43 (0.42) | -0.10 (0.26)
  Week 8 (n=26,25,27,23,24) | -0.36 (0.58) | -0.32 (0.49) | -0.45 (0.31) | -0.52 (0.44) | 0.03 (0.40)
  Week 12 (n=26,24,24,21,24) | -0.38 (0.55) | -0.41 (0.46) | -0.49 (0.35) | -0.57 (0.46) | -0.05 (0.43)

18. Secondary Outcome: C-Reactive Protein (CRP)
Description: The test for CRP is a laboratory measurement for evaluation of an acute phase reactant of inflammation through the use of an ultrasensitive assay. Normal range of CRP is 0 milligram per liter (mg/L) to 10 mg/L. A decrease in the level of CRP indicates reduction in inflammation and therefore improvement.
Time Frame: Baseline, Week 1, 2, 4, 8, 12/EOT
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | CP-690,550 1 mg | CP-690,550 3 mg | CP-690,550 5 mg | CP-690,550 10 mg | Placebo
Number analyzed (Participants) | 28 | 27 | 27 | 26 | 28
mg/L
  Baseline (n=28,27,27,26,28) | 26.71 (31.02) | 27.63 (26.00) | 16.59 (16.15) | 20.03 (21.22) | 22.25 (25.05)
  Week 1 (n=28,26,27,26,28) | 15.45 (21.23) | 13.22 (16.89) | 4.52 (6.49) | 3.29 (4.91) | 20.63 (22.24)
  Week 2 (n=27,27,27,25,26) | 15.79 (20.73) | 10.34 (14.03) | 3.16 (5.37) | 2.15 (3.43) | 18.12 (21.97)
  Week 4 (n=27,26,27,24,25) | 14.33 (21.04) | 9.59 (14.22) | 2.35 (3.36) | 2.40 (5.13) | 17.24 (18.87)
  Week 8 (n=26,25,27,23,24) | 13.82 (22.16) | 4.19 (5.31) | 4.18 (12.36) | 10.72 (23.02) | 15.29 (16.50)
  Week 12 (n=26,24,24,21,24) | 12.04 (21.23) | 8.78 (17.44) | 2.98 (8.72) | 7.00 (16.05) | 17.37 (25.30)

19. Secondary Outcome: Change From Baseline in C-Reactive Protein (CRP) at Week 1, 2, 4, 8 and 12/EOT
Description: as for outcome 18
Time Frame: Baseline, Week 1, 2, 4, 8, 12/EOT
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | CP-690,550 1 mg | CP-690,550 3 mg | CP-690,550 5 mg | CP-690,550 10 mg | Placebo
Number analyzed (Participants) | 28 | 27 | 27 | 26 | 28
mg/L
  Week 1 (n=28,26,27,26,28) | -11.26 (14.29) | -15.37 (20.41) | -12.07 (11.50) | -16.75 (19.28) | -1.62 (11.47)
  Week 2 (n=27,27,27,25,26) | -11.83 (16.03) | -17.29 (20.63) | -13.43 (12.71) | -18.54 (21.03) | -2.38 (16.85)
  Week 4 (n=27,26,27,24,25) | -13.29 (20.00) | -18.35 (22.09) | -14.24 (13.90) | -17.31 (21.16) | -3.26 (16.48)
  Week 8 (n=26,25,27,23,24) | -14.66 (22.72) | -22.90 (24.20) | -12.41 (16.40) | -9.19 (23.29) | -5.83 (16.73)
  Week 12 (n=26,24,24,21,24) | -16.43 (27.15) | -17.89 (28.20) | -10.49 (14.72) | -14.10 (22.34) | -3.75 (19.97)

20. Secondary Outcome: Numeric Index of American College of Rheumatology Response (ACR-n)
Description: ACR-n = calculated for each participant by taking the lowest percentage improvement in (1) SJC or (2) TJC or (3) the median of the remaining 5 components of the ACR response (participant's assessment of disease activity; participant's global assessment of pain; physician's assessment of disease activity; participant's assessment of physical function; an acute phase reactant value - CRP). Negative numbers indicate worsening.
Time Frame: Week 1, 2, 4, 8, 12/EOT
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CP-690,550 1 mg | CP-690,550 3 mg | CP-690,550 5 mg | CP-690,550 10 mg | Placebo
Number analyzed (Participants) | 28 | 27 | 27 | 26 | 28
units on a scale
  Week 1 | 4.80 (32.73) | 6.06 (20.00) | 10.60 (19.13) | 10.73 (42.87) | -11.08 (21.61)
  Week 2 | 8.74 (28.66) | 17.43 (25.30) | 30.61 (26.21) | 25.15 (28.64) | -8.84 (26.69)
  Week 4 | 14.67 (38.45) | 23.83 (32.99) | 40.88 (26.07) | 37.08 (25.42) | -23.54 (51.98)
  Week 8 | 30.40 (33.10) | 31.64 (33.87) | 56.76 (24.53) | 45.62 (29.46) | -18.74 (62.37)
  Week 12 | 30.26 (35.83) | 34.64 (48.37) | 60.16 (24.26) | 52.08 (32.22) | -11.19 (38.76)

21. Secondary Outcome: Area Under the Numeric Index of American College of Rheumatology Response (ACR-n) Curve
Description: ACR-n = calculated for each participant by taking lowest percentage improvement in (1) swollen joint count or (2) tender joint count or (3) the median of remaining 5 components of ACR response (participant's assessment of disease activity; participant's global assessment of pain; physician's assessment of disease activity; participant's assessment of physical function; an acute phase reactant value - CRP). Negative numbers indicate worsening. The AUC for ACR-n is measure of the area under the curve of the mean change from baseline in ACR-n. The trapezoidal rule was used to compute AUC.
Time Frame: Baseline up to Week 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale*weeks
Arm/Group | CP-690,550 1 mg | CP-690,550 3 mg | CP-690,550 5 mg | CP-690,550 10 mg | Placebo
Number analyzed (Participants) | 28 | 27 | 27 | 26 | 28
units on a scale*weeks | 1708.31 (2458.38) | 2096.79 (2355.96) | 3685.71 (1721.44) | 3124.40 (2011.19) | -1346.24 (2995.11)

22. Secondary Outcome: Disease Activity Score Based on 28-Joints Count and C-Reactive Protein (3 Variables) (DAS28-3 [CRP])
Description: DAS28-3 (CRP) was calculated from SJC and TJC using 28 joint count and CRP (mg/L). Total score range: 0 to 9.4, higher score indicated more disease activity. DAS28-3 (CRP) less than or equal to (=<) 3.2 implied low disease activity, >3.2 to 5.1 implied moderate to high disease activity and <2.6 implied remission.
Time Frame: Baseline, Week 1, 2, 4, 8, 12/EOT
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CP-690,550 1 mg | CP-690,550 3 mg | CP-690,550 5 mg | CP-690,550 10 mg | Placebo
Number analyzed (Participants) | 28 | 27 | 27 | 26 | 28
units on a scale
  Baseline (n=28,27,27,26,28) | 5.03 (0.68) | 5.13 (0.94) | 5.00 (0.96) | 4.94 (1.01) | 4.90 (0.87)
  Week 1 (n=28,26,27,26,28) | 4.30 (0.86) | 4.30 (1.10) | 4.09 (1.28) | 3.74 (0.93) | 4.61 (1.08)
  Week 2 (n=27,27,27,25,26) | 4.23 (0.95) | 3.95 (1.18) | 3.46 (1.25) | 3.25 (1.01) | 4.43 (1.11)
  Week 4 (n=27,26,27,24,25) | 3.96 (1.13) | 3.63 (1.05) | 3.21 (1.27) | 2.80 (0.94) | 4.56 (1.15)
  Week 8 (n=26,25,26,23,24) | 3.43 (1.03) | 3.03 (1.10) | 2.77 (0.97) | 2.52 (0.96) | 4.31 (1.21)
  Week 12 (n=26,24,24,21,24) | 3.21 (1.05) | 3.14 (1.27) | 2.55 (0.90) | 2.14 (0.61) | 4.15 (1.36)

23. Secondary Outcome: Disease Activity Score Using 28-Joint Count and Erythrocyte Sedimentation Rate (4 Variables) (DAS28-4 [ESR])
Description: DAS28-4 (ESR) calculated from SJC and TJC using 28 joint count, erythrocyte sedimentation rate (ESR) (millimeters per hour [mm/hour]) and patient's global assessment (PtGA) of disease activity (transformed score ranging 0 to 10; higher score indicated greater affectation due to disease activity). Total score range:0 to 9.4, higher score indicated more disease activity. DAS28-4 (ESR) less than or equal to (=<) 3.2 implied low disease activity, greater than (>) 3.2 to 5.1 implied moderate to high disease activity and less than (<) 2.6=remission.
Time Frame: Baseline, Week 1, 2, 4, 8, 12/EOT
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CP-690,550 1 mg | CP-690,550 3 mg | CP-690,550 5 mg | CP-690,550 10 mg | Placebo
Number analyzed (Participants) | 28 | 27 | 27 | 26 | 28
units on a scale
  Baseline (n=28,27,27,26,28) | 6.11 (0.79) | 6.06 (1.04) | 6.02 (1.03) | 5.86 (0.95) | 5.86 (0.96)
  Week 1 (n=28,26,27,26,28) | 5.42 (0.98) | 5.33 (1.22) | 5.09 (1.34) | 4.88 (1.08) | 5.46 (1.11)
  Week 2 (n=27,27,27,25,26) | 5.29 (1.07) | 5.03 (1.36) | 4.48 (1.37) | 4.28 (1.04) | 5.34 (1.24)
  Week 4 (n=27,26,27,24,25) | 5.00 (1.04) | 4.54 (1.29) | 4.03 (1.43) | 3.72 (1.13) | 5.49 (1.29)
  Week 8 (n=26,25,26,23,24) | 4.37 (1.05) | 4.00 (1.34) | 3.49 (1.21) | 3.13 (1.12) | 5.22 (1.42)
  Week 12 (n=26,24,24,21,24) | 4.07 (0.99) | 3.90 (1.36) | 3.13 (0.99) | 2.83 (0.99) | 5.07 (1.47)

24. Secondary Outcome: 36-Item Short-Form Health Survey (SF-36)
Description: SF-36 is a standardized survey evaluating 8 aspects of functional health and well being: physical and social functioning, physical and emotional role limitations, bodily pain, general health, vitality, mental health. The score for a section is an average of the individual question scores, which are scaled 0-100 (100=highest level of functioning).
Time Frame: Baseline, Week 12/EOT
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CP-690,550 1 mg | CP-690,550 3 mg | CP-690,550 5 mg | CP-690,550 10 mg | Placebo
Number analyzed (Participants) | 28 | 27 | 27 | 26 | 28
units on a scale
  Baseline:Physical functioning (n=28,27,27,26,28) | 37.87 (9.10) | 37.94 (9.37) | 38.87 (10.41) | 40.93 (9.47) | 38.69 (9.80)
  Baseline:Role Physical (n=28,27,27,26,28) | 39.27 (11.83) | 41.43 (13.22) | 44.25 (10.25) | 45.64 (13.33) | 42.77 (11.69)
  Baseline:Bodily Pain (n=28,27,27,26,28) | 37.27 (7.89) | 36.89 (7.53) | 38.59 (8.44) | 40.58 (7.00) | 36.81 (9.61)
  Baseline:General Health (n=28,27,27,26,28) | 37.54 (6.14) | 37.56 (7.53) | 37.57 (10.16) | 38.87 (8.25) | 37.42 (7.00)
  Baseline:Vitality (n=28,27,27,26,28) | 45.07 (11.58) | 46.31 (10.49) | 46.19 (11.13) | 46.69 (9.86) | 46.96 (9.58)
  Baseline:Social Functioning (n=28,27,27,26,28) | 46.72 (13.5) | 42.71 (13.21) | 45.54 (10.47) | 46.78 (11.82) | 45.16 (12.74)
  Baseline:Role-Emotional (n=28,27,27,26,28) | 40.61 (13.00) | 41.05 (13.47) | 45.37 (10.33) | 45.11 (14.93) | 44.91 (13.13)
  Baseline:Mental Health (n=28,27,27,26,28) | 43.07 (10.15) | 44.27 (9.12) | 43.65 (10.11) | 46.97 (10.98) | 45.08 (11.81)
  Baseline:Physical Component (n=28,27,27,26,28) | 37.16 (7.71) | 37.54 (7.92) | 38.75 (8.59) | 40.39 (7.02) | 37.35 (8.56)
  Baseline:Mental Component (n=28,27,27,26,28) | 46.06 (12.16) | 45.81 (11.86) | 47.38 (9.60) | 48.48 (11.72) | 48.36 (12.08)
  Week 12:Physical functioning (n=26,24,24,21,24) | 42.71 (10.07) | 43.27 (9.69) | 46.42 (9.00) | 47.51 (9.86) | 40.72 (9.40)
  Week 12:Role Physical (n=26,24,24,21,24) | 44.61 (10.39) | 46.96 (10.60) | 50.73 (7.19) | 50.32 (9.37) | 44.81 (10.21)
  Week 12:Bodily Pain (n=26,24,24,21,24) | 42.81 (7.05) | 44.58 (8.93) | 48.70 (7.20) | 49.94 (8.45) | 39.77 (7.98)
  Week 12:General Health (n=26,24,24,21,24) | 42.08 (7.07) | 43.14 (8.63) | 45.03 (7.76) | 45.19 (8.06) | 37.78 (8.03)
  Week 12:Vitality (n=26,24,24,21,24) | 50.53 (10.27) | 49.88 (11.52) | 53.65 (11.24) | 52.24 (11.53) | 48.71 (11.20)
  Week 12:Social Functioning (n=26,24,24,21,24) | 48.46 (10.37) | 46.62 (12.49) | 51.85 (7.36) | 52.43 (8.20) | 47.99 (12.12)
  Week 12:Role-Emotional (n=26,24,24,21,24) | 47.51 (8.64) | 46.16 (12.08) | 47.78 (10.12) | 48.47 (9.83) | 44.70 (12.15)
  Week 12:Mental Health (n=26,24,24,21,24) | 50.22 (7.96) | 47.90 (11.87) | 51.53 (7.33) | 49.07 (12.51) | 46.25 (13.81)
  Week 12:Physical Component (n=26,24,24,21,24) | 41.21 (9.42) | 43.87 (7.75) | 47.27 (6.61) | 48.39 (7.18) | 39.77 (6.59)
  Week 12:Mental Component (n=26,24,24,21,24) | 51.90 (8.68) | 48.93 (13.44) | 52.07 (8.99) | 50.68 (10.10) | 49.00 (13.09)

25. Secondary Outcome: Euro Quality of Life (EQ-5D)- Health State Profile Utility Score
Description: EQ-5D: participant rated questionnaire to assess health-related quality of life in terms of a single utility score. Health State Profile component assesses level of current health for 5 domains: mobility, selfcare, usual activities, pain and discomfort, and anxiety and depression; 1 indicates better health state (no problems); 3 indicates worst health state (confined to bed). Scoring formula developed by EuroQoL Group assigns a utility value for each domain in the profile. Score is transformed and results in a total score range -0.594 to 1.000; higher score indicates a better health state.
Time Frame: Baseline, Week 12/EOT
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CP-690,550 1 mg | CP-690,550 3 mg | CP-690,550 5 mg | CP-690,550 10 mg | Placebo
Number analyzed (Participants) | 28 | 27 | 27 | 26 | 28
units on a scale
  Baseline (n=28,27,27,26,28) | 0.55 (0.26) | 0.45 (0.29) | 0.58 (0.24) | 0.55 (0.32) | 0.51 (0.33)
  Week 12 (n=26,24,24,21,24) | 0.65 (0.23) | 0.70 (0.27) | 0.79 (0.13) | 0.78 (0.28) | 0.59 (0.27)

26. Secondary Outcome: Medical Outcome Study- Sleep Scale (MOS-SS)
Description: Participant-rated 12 item questionnaire assess constructs of sleep over past week.7 subscales:sleep disturbance(SD),snoring(Sno),awakened short of breath(ASOB),sleep adequacy(Ade),somnolence(Som)(range:0-100);sleep quantity(Qua)(range:0-24),optimal(Opt) sleep(yes:1,no:0),9 item index measures of sleep disturbance provide composite scores:sleep problem summary(SPS),overall SP(OSP).Except Ade,Opt,Qua,higher scores=more impairment.Scores transformed(actual raw score(RS) minus lowest possible score divided by possible RS range*100);total score range:0-100;higher score=more intensity of attribute.
Time Frame: Baseline, Week 2, 12/EOT
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CP-690,550 1 mg | CP-690,550 3 mg | CP-690,550 5 mg | CP-690,550 10 mg | Placebo
Number analyzed (Participants) | 28 | 27 | 27 | 26 | 28
units on a scale
  Baseline: SPS (n=28,27,27,26,28) | 27.38 (11.42) | 27.41 (14.36) | 29.38 (17.54) | 30.51 (18.78) | 23.93 (12.57)
  Baseline: OSP (n=28,27,27,26,28) | 28.00 (10.53) | 27.55 (12.40) | 31.07 (17.38) | 31.28 (18.60) | 25.95 (12.89)
  Baseline: Ade (n=28,27,27,26,28) | 52.86 (24.47) | 52.96 (24.93) | 49.63 (27.80) | 51.54 (26.64) | 58.57 (27.98)
  Baseline: ASOB (n=28,27,27,26,28) | 3.57 (9.51) | 4.44 (10.13) | 8.15 (22.37) | 10.00 (14.14) | 3.57 (7.80)
  Baseline: SD (n=28,27,27,26,28) | 24.06 (17.70) | 23.84 (21.10) | 25.28 (20.95) | 25.77 (21.45) | 21.43 (16.66)
  Baseline: Opt (n=28,27,27,26,28) | 0.61 (0.50) | 0.30 (0.47) | 0.41 (0.50) | 0.42 (0.50) | 0.39 (0.50)
  Baseline: Qua (n=28,27,27,26,28) | 6.61 (1.10) | 6.37 (1.45) | 6.30 (0.87) | 6.38 (1.27) | 6.43 (1.29)
  Baseline: Sno (n=28,27,27,26,28) | 25.00 (27.01) | 32.59 (34.26) | 31.85 (31.99) | 23.08 (29.77) | 31.43 (29.53)
  Baseline: Som (n=28,27,27,26,28) | 29.05 (19.13) | 28.64 (17.81) | 34.57 (25.22) | 32.05 (22.86) | 31.90 (19.49)
  Week 2: SPS (n=27,27,27,25,26) | 27.04 (11.52) | 25.19 (12.55) | 22.10 (16.28) | 27.87 (19.41) | 26.67 (16.49)
  Week 2: OSP (n=28,27,27,26,28) | 27.61 (10.05) | 25.62 (12.35) | 22.78 (15.29) | 27.47 (18.67) | 27.74 (15.79)
  Week 2: Ade (n=28,27,27,26,28) | 53.33 (23.86) | 54.81 (22.42) | 64.07 (27.49) | 51.20 (29.48) | 55.38 (25.33)
  Week 2: ASOB (n=28,27,27,26,28) | 5.93 (16.47) | 4.44 (8.47) | 8.15 (20.95) | 7.20 (12.75) | 4.62 (11.74)
  Week 2: SD (n=28,27,27,26,28) | 22.31 (14.11) | 19.68 (19.19) | 17.92 (14.88) | 21.40 (21.39) | 21.44 (18.22)
  Week 2: Opt (n=28,27,27,26,28) | 0.63 (0.49) | 0.44 (0.51) | 0.56 (0.51) | 0.52 (0.51) | 0.38 (0.50)
  Week 2: Qua (n=28,27,27,26,28) | 6.70 (0.82) | 6.52 (1.16) | 6.70 (1.14) | 6.84 (1.25) | 6.50 (1.24)
  Week 2: Sno (n=28,27,27,26,28) | 25.19 (26.94) | 25.19 (22.60) | 23.70 (29.89) | 17.60 (24.71) | 30.00 (34.06)
  Week 2: Som (n=28,27,27,26,28) | 30.37 (18.05) | 29.14 (19.93) | 27.90 (23.46) | 26.13 (23.88) | 35.64 (20.65)
  Week 12: SPS (n=26,24,24,21,24) | 24.49 (10.83) | 24.17 (14.22) | 23.89 (11.78) | 25.56 (14.47) | 28.75 (14.24)
  Week 12: OSP (n=26,24,24,21,24) | 25.19 (10.33) | 24.19 (13.39) | 23.08 (10.74) | 24.52 (14.29) | 29.56 (13.10)
  Week 12: Ade (n=26,24,24,21,24) | 60.00 (22.63) | 58.75 (26.75) | 51.67 (24.08) | 53.33 (23.94) | 54.17 (19.54)
  Week 12: ASOB (n=26,24,24,21,24) | 6.92 (13.79) | 9.17 (14.42) | 5.00 (10.63) | 3.81 (8.05) | 10.00 (20.43)
  Week 12: SD (n=26,24,24,21,24) | 20.34 (13.42) | 19.22 (18.43) | 14.43 (10.52) | 18.99 (19.05) | 21.09 (16.56)
  Week 12: Opt (n=26,24,24,21,24) | 0.54 (0.51) | 0.38 (0.49) | 0.38 (0.49) | 0.48 (0.51) | 0.46 (0.51)
  Week 12: Qua (n=26,24,24,21,24) | 6.35 (1.20) | 6.54 (1.28) | 6.38 (0.97) | 6.71 (1.38) | 6.54 (1.53)
  Week 12: Sno (n=26,24,24,21,24) | 24.62 (22.13) | 21.67 (22.78) | 29.17 (32.83) | 13.33 (20.33) | 33.33 (31.02)
  Week 12: Som (n=26,24,24,21,24) | 30.26 (18.59) | 25.28 (20.99) | 25.28 (16.33) | 24.13 (23.24) | 40.28 (19.51)

27. Secondary Outcome: Functional Assessment of Chronic Illness Therapy (FACIT)-Fatigue Scale
Description: FACIT-F is a 13-item questionnaire. Participant scored each item on a 5-point scale: 0 (Not at all) to 4 (Very much). The larger the participant's response to the questions (with the exception of 2 negatively stated), the greater the fatigue. For all questions, except for the 2 negatively stated ones, the code was reversed and a new score was calculated as 4 minus the participant's response. The sum of all responses resulted in the FACIT-Fatigue score for a total possible score of 0 (worse score) to 52 (better score). A higher score reflected an improvement in the participant's health status.
Time Frame: Baseline, Week 2, 12/EOT
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CP-690,550 1 mg | CP-690,550 3 mg | CP-690,550 5 mg | CP-690,550 10 mg | Placebo
Number analyzed (Participants) | 28 | 27 | 27 | 26 | 28
units on a scale
  Baseline (n=28,27,27,26,28) | 34.25 (10.45) | 33.37 (11.03) | 34.48 (9.99) | 36.85 (9.43) | 37.07 (9.87)
  Week 2 (n=27,27,27,25,26) | 36.78 (8.64) | 36.48 (9.72) | 39.30 (10.56) | 40.80 (6.87) | 37.38 (10.31)
  Week 12 (n=26,24,24,21,24) | 39.35 (7.47) | 37.96 (9.95) | 42.79 (8.47) | 40.76 (10.65) | 36.46 (9.93)

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | CP-690,550 1 mg | CP-690,550 3 mg | CP-690,550 5 mg | CP-690,550 10 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 1/28 | 1/27 | 1/27 | 2/26 | 0/28
Other Adverse Events (participants affected / at risk) | 14/28 | 16/27 | 19/27 | 19/26 | 11/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CP-690,550 1 mg (N=28) | CP-690,550 3 mg (N=27) | CP-690,550 5 mg (N=27) | CP-690,550 10 mg (N=26) | Placebo (N=28)
Cardiac failure (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Foot deformity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | CP-690,550 1 mg (N=28) | CP-690,550 3 mg (N=27) | CP-690,550 5 mg (N=27) | CP-690,550 10 mg (N=26) | Placebo (N=28)
Cataract (Eye disorders) | 0 | 0 | 0 | 1 | 0
Conjunctivitis (Eye disorders) | 0 | 0 | 0 | 0 | 1
Dry eye (Eye disorders) | 0 | 0 | 0 | 1 | 0
Eyelid pain (Eye disorders) | 0 | 0 | 1 | 0 | 0
Vision blurred (Eye disorders) | 0 | 0 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 1 | 1 | 0
Gastric mucosal lesion (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Paraesthesia oral (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Stomach discomfort (Gastrointestinal disorders) | 0 | 0 | 3 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 1 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 1 | 0
Malaise (General disorders) | 1 | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 1 | 0 | 0 | 0
Acute tonsillitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Cystitis (Infections and infestations) | 0 | 0 | 1 | 1 | 0
Dermatitis infected (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Enterocolitis viral (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Erysipelas (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 2 | 0 | 1 | 1
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Localised infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 3 | 1 | 1 | 4 | 4
Paronychia (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Peritonsillitis (Vascular disorders) | 0 | 0 | 0 | 1 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 2 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 1 | 0
Tinea pedis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 1
Viral upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Vulvovaginal candidiasis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Vulvovaginitis trichomonal (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 1 | 1
Foot fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Joint sprain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Thermal burn (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 1 | 2 | 6 | 2 | 1
Apolipoprotein A-I increased (Investigations) | 0 | 1 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 2 | 4 | 1 | 1
Blood alkaline phosphatase increased (Investigations) | 0 | 1 | 0 | 0 | 0
Blood cholesterol increased (Investigations) | 0 | 3 | 1 | 1 | 0
Blood creatine phosphokinase MM increased (Investigations) | 0 | 0 | 1 | 0 | 0
Blood triglycerides increased (Investigations) | 1 | 1 | 1 | 2 | 0
Epstein-Barr virus test positive (Investigations) | 1 | 0 | 0 | 0 | 0
Haemoglobin decreased (Investigations) | 0 | 0 | 1 | 0 | 0
Low density lipoprotein increased (Investigations) | 0 | 2 | 1 | 2 | 0
Lymphocyte count decreased (Investigations) | 0 | 1 | 0 | 0 | 0
Lymphocyte percentage decreased (Investigations) | 0 | 1 | 1 | 0 | 0
Viral DNA test positive (Investigations) | 0 | 1 | 0 | 0 | 0
White blood cell count decreased (Investigations) | 0 | 0 | 2 | 1 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Monarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Muscle fatigue (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Muscle tightness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Cervical myelopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 2 | 0 | 2 | 0 | 1
Hypoaesthesia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Sciatica (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1
Calculus ureteric (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
Cystitis-like symptom (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Enuresis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Breast pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0
Metrorrhagia (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 2
Haemorrhage subcutaneous (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Purpura (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 0 | 1 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 2 | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.